CLINICAL TRIAL: NCT01016639
Title: Phase I-II Study of Capecitabine and Oxaliplatin in Combination With Radiotherapy in Patients With Unresectable Gastro-Intestinal Cancer
Brief Title: Study of Capecitabine and Oxaliplatin in Combination With Radiotherapy in Patients With Unresectable Gastro-Intestinal Cancer
Acronym: CORGI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Roche Pharma AG (Industry); Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version1
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Stomach Cancer; Gall Bladder Cancer; Bile Ductus Cancer; Pancreas Cancer; Colorectal Cancer
Keywords: Stomach cancer; Gall bladder cancer; Bile ductus cancer; Pancreas cancer; Colorectal cancer; Chemo radiotherapy; Phase I-II; Oxaliplatin; Capecitabine; Response
MeSH Terms: conditions — Stomach Neoplasms; Gallbladder Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemoradiotherapy (Experimental)
  Interventions: Other: oxaliplatin, capecitabine, radiotherapy

INTERVENTIONS:
Other: oxaliplatin, capecitabine, radiotherapy

SUMMARY:
The purpose with this study is to evaluate treatment with radio chemotherapy (oxaliplatin and capecitabine) given concommitant with radiotherapy in patients with gastrointestinal tumors. The trial consists ot two separate studies; CORGI-U in patients with stomach- bile ducts- gallbladder and pancreas cancer, and CORGI-L in patients with colorectal cancer.

CORGI-U will be designed as a phase-I-II-study,in which the first part will be a chemotherapy dose finding study, followed by a phase II part to establish response rates. All subjects receives radiotherapy concommitant.

CORGI-L is a phase II trial, in which patients are treated with chemotherapy at fixed doses with radiotherapy concommitant.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Measurable disease according to RECIST
* ECOG Performance Status 0-1
* ANC over 1.5 x 10 9/L
* Platelets over 100 x 10 9/L
* Creatinine less than 1.5 x ULN
* Bilirubin less than 1.5 x ULN
* ALT less than 2.5 x ULN
* Signed informed concent

Exclusion Criteria:

* Prior radiotherapy to the same local
* Prior chemotherapy for locally advanced or metastatic disease
* Pregnancy or breast feeding
* Peripheral neuropathy more than grade 1
* Uncontrolled diarrhéa
* Other serious uncontrolled concomitant illness
* Lymph node metastasis that can not be included in the GTV (gross tumor volume), without exceeding the stipulated radiotherapy doses in organs at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2003-06; Primary Completion 2007-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Johnsson, MD, PhD, Principal Investigator — University Hospital Lund
Locations (5):
- Sweden (5):
  - Centralsjukhuset, Dept of Oncology, Karlstad
  - University Hospital Lund, Lund
  - University Hospital Malmö, Dept of Oncology, Malmo
  - Karolinska University Hospital, Stockholm
  - Akademiska Sjukhuset, Uppsala